CLINICAL TRIAL: NCT05073575
Title: Healing of Periodontal Suprabony Defects Following Treatment With Open Flap Debridement With or Without Hyaluronic Acid (HA) Application
Brief Title: Application of Hyaluronic Acid in the Treatment of Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luca Ramaglia, Clinical Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 235/21
Record Dates: First submitted 2021-09-06; First posted 2021-10-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Bone Loss
Keywords: Hyaluronic Acid; Suprabony Defect; Surgical Periodontal Therapy; Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: The study will be designed as a double-arm randomized controlled clinical trial. The suprabony defects of subjects allocated in HA group will be treated with open flap debridement and application of hyaluronic acid, while the suprabony defects of No-HA Group will be treated with open flap debridement alone. The null hypothesis of no statistically significant differences between the two modalities for the treatment of suprabony defects will be tested.
Who Masked: Participant
Masking Description: Only patients will be unaware of the type of treatment performed, with prior written informed consent. So, they will be divided in the two groups of study after a process of randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid Group (Experimental): Hyaluronic acid gel will be applied to exposed dental roots surfaces, after scaling and root planing therapy
  Interventions: Procedure: Hyaluronic acid
- No-hyaluronic acid Group (Active Comparator): Only scaling and root planning will be performed on the exposed dental roots surfaces
  Interventions: Procedure: No-hyaluronic acid

INTERVENTIONS:
Procedure: Hyaluronic acid — After local anesthesia, an access flap will be prepared. Scaling and root planning will be performed combining the use of metal curettes and power-driven instrumentation by means of ultrasonic scaler.
  Hyaluronic acid gel will be applied to exposed roots surface, followed by a tension-free primary closure of the surgery wound by means of 5-0 monofilament (polypropylene) non-resorbable suturing material.
  Arms: Hyaluronic acid Group
Procedure: No-hyaluronic acid — An access flap will be prepared in order to perform scaling and root planning therapy with the use of metal curettes.
  After intervention, a tension-free primary closure of the interdental papillae and of the mucoperiosteal flaps by means of 5-0 monofilament (polypropylene) non-resorbable suturing materia will be performed
  Arms: No-hyaluronic acid Group

SUMMARY:
The aim of the present investigation will be evaluated the healing of suprabony defects following surgical flap elevation and hyaluronic acid application respect to surgical flap elevation alone.

A total of 80 patients will be enrolled, selected by inclusion and exclusion criteria and randomly divided in two groups: hyaluronic acid group and no-hyaluronic acid group.

DETAILED DESCRIPTION:
The objective of the study will be compare the healing of suprabony defects following treatment with either open flap debridement (OFD) and application of hyaluronic acid (HA) with OFD alone.

Eighty patients with suprabony periodontal defects will be randomly assigned to treatment with open flap debridement and application of hyaluronic acid (HA Group) or open flap debridement alone (No-HA Group).

Primary outcome will be Clinical Attachment Level (CAL) gain, while the secondary outcomes will be Probing Depth (PD) and Gingival Recession (GR).

After local anesthesia, an access flap will be prepared. Depending on the mesiodistal width of the interproximal space, two different incision techniques will be selected to access the suprabony defect area. The modified papilla preservation technique (MMPT) will be used at sites with an interproximal width > 2 mm, whereas the simplified papilla preservation technique (SPPT) will be applied at sites with an interproximal width ≤ 2 mm. Then, a mucoperiosteal flap will be reflected.

Scaling and root planning will be performed combining the use of metal curettes and power-driven instrumentation by means of ultrasonic scaler.

Hyaluronic acid will be applied to exposed roots surface only in HA Group followed, for both groups, by a tension-free primary closure of the interdental papillae and of the mucoperiostal flaps by means of 5-0 monofilament (polypropylene) non-resorbable suturing material.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with periodontitis
* Age ≥ 18 years old
* Single-rooted and multi-rooted teeth
* Presence of suprabony periodontal defects at a minimum of two adjacent teeth and a maximum of 7 adjacent teeth in either the maxilla or the mandible with a PD ≥ 5 mm after completion of non-surgical periodontal treatment and re-evaluation
* Intrabony defect with an intraosseous component < 2 mm

Exclusion Criteria:

* Patients with systemic diseases
* Prolonged antibiotic or anti-inflammatory treatment within 4 weeks prior to surgery
* Pregnant or lactating
* Tobacco smokers (≥ 10 cigarettes per day)
* Multi-rooted teeth with furcation involvement
* Increased tooth mobility (grade II and III)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of Clinical Attachment Level (CAL) gain (millimeters) | baseline, 6 months after surgical periodontal therapy
  Distance from the cementoenamel junction to the bottom of the pocket

SECONDARY OUTCOMES:
Change of Probing Depth (PD) (millimeters) | baseline, 6 months after surgical periodontal therapy
  Distance from the gingival margin to the bottom of the pocket
Change of Gingival Recession (GR) (millimeters) | baseline, 6 months after surgical periodontal therapy
  Distance from gingival margin to the cementoenamel junction

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No